CLINICAL TRIAL: NCT02968225
Title: Using Serious Game Technology to Improve Sensitivity to Eye Gaze in Autism
Acronym: SAGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, K. Suzanne Scherf, Associate Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R61MH110624 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants randomized into intervention or standard care control conditions
Who Masked: Participant, Investigator
Masking Description: Given the design of the study, parents and adolescents will know the condition to which they have been assigned. However, researchers involved in data collection will be blinded from condition assignment during the pre-intervention data collection session as these data will be collected prior to randomization. Also, the research team is not involved in the randomization process. The research team members who are involved in ensuring the fidelity of the intervention are not involved in data collection procedures. Although we will attempt to limit unblinding, it is not possible for researchers involved in data collection to be completely blinded to the assignment of participant condition at the post-intervention visit as we cannot prohibit participants from talking to researchers about their experience in the study. Importantly, the primary outcome measures are believed to be robust to investigator bias.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer Game (Experimental): All Computer Game participants will complete:
  * online screening
  * Diagnostic and eye-tracking pre-testing
  * 2 month intervention
  * Eye-tracking post-testing
  Interventions: Behavioral: Computer Game
- Waitlist control (No Intervention): All Treatment as usual control participants will complete:
  * online screening
  * Diagnostic and eye-tracking pre-testing
  * Eye-tracking post-testing

INTERVENTIONS:
Behavioral: Computer Game — The game involves viewing subtle nonverbal behaviors of game characters for the purpose of executing their own goal-directed behavior in the game related to solving various crimes. The learning involves interpreting nonverbal cues on the animated characters, such as pointing, head turns, eye gaze cues.
  Arms: Computer Game

SUMMARY:
The investigators hypothesize that this serious game (designed to provide a learning environment that maximizes opportunities for adolescents with autism to discover the functional utility of eye gaze) will improve sensitivity to eye gaze cues, specifically to identify gazed-at objects, and will also lead to increased social attention to faces in adolescents with autism. The investigators will test this hypothesis in a small-scale exploratory randomized control trial that will include both behavioral and eye tracking outcome measures.

ELIGIBILITY:
Inclusion criteria:

1. parent/caregiver of an adolescent with a diagnosis of ASD,
2. parent/caregiver and adolescent with ASD both native English speakers,
3. adolescent with ASD aged between 10-18 years at enrollment,
4. adolescent has normal vision and hearing with correction as indicated by parent report,
5. adolescent is able to use a computer for the purposes of game play,
6. adolescent scores > 80% correct (i.e., 0.5 SD less than M of TD adolescents) on online eye gaze screening task,
7. ASD diagnosis of adolescent confirmed in lab via the Autism Diagnostic Observation Schedule,
8. Full Scale IQ of adolescent determined to be between 70-130 on the Kaufman Brief Intelligence Test,
9. reading ability of adolescent determined to be at least a second grade level as assessed by the Oral and Written Language Scales,
10. adolescent is capable of cooperating with testing,
11. parent/caregiver and adolescent both consent/assent to participate in the research.

Exclusion Criteria

1. adolescent has had seizures within the previous two years,
2. family lacks stable home internet,
3. parent or adolescent refuses to consent/assent to take part in the research,
4. adolescent is 18 and has a legal guardian, prohibiting him/her from legally consenting, or
5. adolescent is 18 and cannot understand the consent (i.e., fails consent quiz).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Static Eye Gaze Following Task | 2 months
  Eye tracking and accuracy
Dynamic Eye Gaze Following Task | 2 Months
  Eye tracking and accuracy
Social/Visual Attention Task | 2 Months
  Eye tracking

SECONDARY OUTCOMES:
Social Responsiveness Scale | 2 months
  Parents completing measure of autism-like behavior in adolescents
Social Skills Inventory System - Child version | 2 months
  Adolescents completing measure of social skills and problem behaviors in themselves
Social Skills Inventory System - Adult version | 2 months
  Parents completing measure of social skills and problem behaviors in adolescents
Treatment as Usual | 2 months
  Parents reporting on social and behavioral treatments adolescents receiving in and out of school

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Scherf, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared in the NIMH National Data Archive
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Scherf KS, Griffin JW, Geier CF, Smyth JM. Social visual attention as a treatment outcome: evaluating the social games for autistic adolescents (SAGA) intervention. Sci Rep. 2024 Jan 5;14(1):619. doi: 10.1038/s41598-024-51332-z. PMID 38182792
- [Derived] Scherf KS, Griffin JW, Judy B, Whyte EM, Geier CF, Elbich D, Smyth JM. Improving sensitivity to eye gaze cues in autism using serious game technology: study protocol for a phase I randomised controlled trial. BMJ Open. 2018 Oct 4;8(9):e023682. doi: 10.1136/bmjopen-2018-023682. PMID 30287612
- See also: Improving sensitivity to eye gaze cues in autism using serious game technology: study protocol for a phase I randomised controlled trial — https://bmjopen.bmj.com/content/bmjopen/8/9/e023682.full.pdf